CLINICAL TRIAL: NCT00991510
Title: Comparative Bioavailability of Myfenax® (Teva) and CellCept® (Roche) in Stable Patients After Renal Transplantation
Brief Title: Comparative Bioavailability of Myfenax® and CellCept® in Kidney Transplant Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment and lack of time to product launch
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 116B8; 2009-010562-31 (EudraCT Number)
Record Dates: First submitted 2009-08-29; First posted 2009-10-08 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: Stable Renal Transplant Recipients
Keywords: renal transplantation; mycophenolate mofetil; pharmacokinetics; immunosuppression
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reference/Test/Test (Experimental): The reference product was CellCept® and test product was Myfenax®. In period I, participants received CellCept on Days 1-14. In period II, participants crossed-over to receive Myfenax on Days 15-28. In period III, participants received Myfenax until the end of the study (Days 29-112).
  Doses of mycophenolate mofetil were at least 500 mg twice daily, morning and evening.
  Interventions: Drug: mycophenolate mofetil (Myfenax); Drug: mycophenolate mofetil (Cellcept)
- Test/Reference/Reference (Experimental): The test product was Myfenax® and the reference product was CellCept®. In period I, participants received Myfenax on Days 1-14. In period II, participants crossed-over to receive CellCept on Days 15-28. In period III, participants received CellCept until the end of the study (Days 29-112).
  Doses of mycophenolate mofetil were at least 500 mg twice daily, morning and evening.
  Interventions: Drug: mycophenolate mofetil (Myfenax); Drug: mycophenolate mofetil (Cellcept)

INTERVENTIONS:
Drug: mycophenolate mofetil (Myfenax) — Each participant received at least 500 mg orally, twice daily (morning and evening) during those study periods labeled as 'T' (test drug). Participants receive the dose equivalent to the pre-study dose (within the recommended therapeutic range) of mycophenolate mofetil.
  Other Names: Myfenax®
Drug: mycophenolate mofetil (Cellcept) — Each participant received at least 500 mg orally, twice daily (morning and evening) during those study periods labeled as 'R' (reference drug). Participants receive the dose equivalent to the pre-study dose (within the recommended therapeutic range) of mycophenolate mofetil.
  Other Names: CellCept®

SUMMARY:
The purpose of the study is to further investigate how much of the drug substance "mycophenolate mofetil" can be found in the blood of patients with kidney or renal transplants when treated with Myfenax® or CellCept®. Additionally, the safety and side effects of the two products will be compared. All information already available on these products indicates that the safety profiles of the two products will be the same.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipients at least 12 months post-transplantation aged ≥ 18 years.
* Maintenance treatment with mycophenolate mofetil (in combination with tacrolimus with or without corticosteroids).
* Stable dose of mycophenolate mofetil (≥ 500 mg twice daily) with no changes in immunosuppressive regimen for at least 6 weeks prior to the start of the study.
* Stable renal graft function for at least 3 months.
* Female patients must be either post-menopausal for ≥ 1 year, be surgically sterilized or a negative pregnancy test will be required immediately prior to study entry and such patients must continue to use effective contraception.
* Willingness to undergo the study-related procedures.
* Ability to comprehend and willingness to sign informed consent form.

Exclusion Criteria:

* History of allergy to mycophenolate mofetil, mycophenolic acid or any of the ingredients.
* Multi-organ recipients (e.g., kidney and pancreas) or previous transplant with any organ other than kidney.
* Rejection within the past 6 months prior to the start of the study.
* Severe clinically relevant co-existing disease.
* History of cancer other than skin cancer that has been cured.
* History of serious clinically relevant digestive system disease during the last 12 months prior to start of the study.
* Known or suspected hereditary deficiency of hypoxanthine-guanine-phosphoribosyltransferase (e.g., Lesch-Nyhan syndrome, Kelley-Seegmiller syndrome).
* Known or suspected liver impairment.
* Clinically significant thrombocytopenia, anaemia, leukopenia, or neutropenia
* Clinically significant laboratory and/or physical changes during the last 2 months prior to the start of the study.
* Use of azathioprine, cholestyramine, sevelamer, or probenecid within 2 weeks prior to the first administration of study medication.
* Change in concomitant medication during the 6 weeks prior to start of the study.
* Use of any drug, prescribed or over-the-counter, (except stable concomitant medication) within 2 weeks prior to the first administration of study medication.
* Planned or expected requirement for the use of live attenuated vaccines during the study.
* Positive testing for HIV, Hepatitis B and C.
* Clinical symptoms or laboratory evidence of cytomegalovirus infection in the last 6 month.
* Pregnant or breast-feeding women.
* Women of childbearing potential unable or unwilling to practice effective contraceptive measures for the duration of the study and for 6 weeks after the end of the study.
* History of known or suspected alcohol or drug abuse.
* Any other condition of the patient that, in the opinion of the investigator may compromise evaluation of the study treatment or may jeopardize patient's compliance or adherence to protocol requirements.
* Previous enrollment in this study or participation in any other drug investigational trial within the past 6 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gere Sunder-Plassman, Prof.,MD, Principal Investigator — Medical University Vienna

REFERENCES:
- [Result] Sunder-Plassmann G et al.: Results of a Comparative Bioavailability Study of Myfenax (Teva) and CellCept (Roche) in Stable Kidney Transplant Recipients. American Transplant Congress 2011. Abstract Number: 250308
- [Result] Sunder-Plassmann G, Reinke P, Rath T, Wiecek A, Nowicki M, Moore R, Lutz J, Gaggl M, Ferkl M. Comparative pharmacokinetic study of two mycophenolate mofetil formulations in stable kidney transplant recipients. Transpl Int. 2012 Jun;25(6):680-6. doi: 10.1111/j.1432-2277.2012.01475.x. Epub 2012 Apr 16. PMID 22500920

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 100 subjects were planned. A total of 47 subjects were screened in the study. Four subjects were not randomised, i.e., two subjects withdrew consent, one subject had a protocol violation, and one subject was a screening failure (did not meet eligibility criteria).
Period: Period I (Days 1-14)
Arm/Group | Reference/Test/Test | Test/Reference/Reference
Started | 22 | 21
Completed | 21 | 21
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Period II (Days 15-28)
Arm/Group | Reference/Test/Test | Test/Reference/Reference
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0
Period: Period III (Days 29-112)
Arm/Group | Reference/Test/Test | Test/Reference/Reference
Started | 21 | 21
Completed | 20 | 20
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reference/Test/Test | Test/Reference/Reference | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (13.73) | 51.7 (13.55) | 50.7 (13.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 11 | 13 | 24
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 1
  Caucasian | 21 | 21 | 42
Height [Mean (Standard Deviation); unit: meters] | 1.711 (0.1061) | 1.718 (0.0983) | 1.714 (0.1012)
Weight [Mean (Standard Deviation); unit: kilograms] | 77.19 (14.856) | 77.23 (15.661) | 77.21 (15.072)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.24 (3.756) | 25.93 (3.422) | 26.09 (3.557)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC(0-6h)) of Mycophenolate Mofetil
Description: Area under the plasma concentration-time curve during a dosage interval at steady state (calculated using the trapezoidal rule, from t = 0 to t = 6 hours).
Time Frame: Day 14 and Day 28 (end of first two cross-over periods) before drug administration and at 30 min, 1 hour, 1.5, 2, 3, 4, 5, 6, 8, 10, and 12 hours after drug administration
Population: PK population. Two participants were excluded from the PK population: one dropped out of the study during the first period so had no PK samples. The other was omitted due to protocol violations.
Measure: Mean (Standard Deviation); unit: hour* µg /ml
Groups:
- CellCept: Timeframes in periods I and II when participants took CellCept in this cross-over study. Doses of mycophenolate mofetil were at least 500 mg twice daily, morning and evening.
- Myfenax: Timeframes in periods I and II when participants took Myfenax in this cross-over study. Doses of mycophenolate mofetil were at least 500 mg twice daily, morning and evening.
Arm/Group | CellCept | Myfenax
Number analyzed (Participants) | 41 | 41
hour* µg /ml | 33.523 (15.1265) | 31.100 (15.4198)
Statistical Analysis 1: Comparison: CellCept vs Myfenax; A total of 100 subjects were planned to be enrolled, allowing for 10% drop-out rate. Based on previous single dose studies, the intra-subject coefficients of variation were 14% and 50% for AUC and Cmax, respectively. Based on the literature similar intra subject coefficients of variation were observed in steady-state patients. With these expected CV(%) and an expected ratio of Cmax within 0.95 and 1.05, the study should have a power of at least 80 % to show bioequivalence with 80 subjects; Test type: Non-Inferiority or Equivalence — Bioequivalence was accepted if the calculated 90 % CIs were within 0.80-1.25; ANOVA; adjusted least-squares mean ratio = 0.923, 90% CI 2-sided [0.865 to 0.984]

2. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC(0-tau)) of Mycophenolate Mofetil
Description: For participants with a 0-12h profile: Area under the plasma concentration-time curve during a dosage interval at steady state (calculated using the trapezoidal rule, from t = 0 to t = 12 hours). For participants with a 0-6h profile: AUC(0-tau) was calculated based on AUC(0-6h) using the extrapolation formula according to Fleming.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour* µg /ml
Arm/Group | CellCept | Myfenax
Number analyzed (Participants) | 41 | 41
hour* µg /ml | 49.846 (20.8278) | 48.255 (21.2246)
Statistical Analysis 1: Comparison: CellCept vs Myfenax; Test type: Non-Inferiority or Equivalence — Bioequivalence was accepted if the calculated 90 % CIs were within 0.80-1.25; ANOVA; adjusted least-squares mean ratio = 0.959, 90% CI 2-sided [0.899 to 1.023]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Mycophenolate Mofetil
Description: Cmax was directly obtained from measured values of plasma concentrations.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg /ml
Arm/Group | CellCept | Myfenax
Number analyzed (Participants) | 41 | 41
µg /ml | 16.189 (9.9448) | 14.308 (8.3432)
Statistical Analysis 1: Comparison: CellCept vs Myfenax; Test type: Non-Inferiority or Equivalence — Bioequivalence was accepted if the calculated 90 % CIs were within 0.80-1.25; ANOVA; adjusted least-squares mean ratio = 0.873, 90% CI 2-sided [0.787 to 0.968]

4. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) of Mycophenolate Mofetil
Description: Cmin was directly obtained from measured values of plasma concentrations.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg /ml
Arm/Group | CellCept | Myfenax
Number analyzed (Participants) | 41 | 41
µg /ml | 1.584 (0.7801) | 1.567 (0.7387)
Statistical Analysis 1: Comparison: CellCept vs Myfenax; Test type: Non-Inferiority or Equivalence — Bioequivalence was accepted if the calculated 90 % CIs were within 0.80-1.25; ANOVA; adjusted least-squares mean ratio = 0.985, 90% CI 2-sided [0.877 to 1.106]

5. Secondary Outcome: Plasma Concentrations of Mycophenolate Mofetil in Pre-Administration Samples (Cpd)
Description: Cpd was directly obtained from measured values of plasma concentrations.
Time Frame: Day 14 and Day 28 (end of first two cross-over periods) before drug administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg /ml
Arm/Group | CellCept | Myfenax
Number analyzed (Participants) | 41 | 41
µg /ml | 2.693 (1.7001) | 3.001 (2.0863)

6. Secondary Outcome: Degree of Fluctuation of the Concentration Levels of Mycophenolate Mofetil Over One Dosing Interval (PTF)
Description: PTF was calculated as: (Cmax-Cmin)/(AUCt/t)*100
Time Frame: Day 14 and Day 28 (end of first two cross-over periods) before drug administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of AUC for a dosing interval
Arm/Group | CellCept | Myfenax
Number analyzed (Participants) | 41 | 41
percentage of AUC for a dosing interval | 351.05 (161.195) | 323.67 (156.018)

7. Secondary Outcome: Time Corresponding to Occurrence of Cmax (Tmax) of Mycophenolate Mofetil
Description: Tmax was directly obtained from measured values.
Time Frame: Day 14 and Day 28 (end of first two cross-over periods) before drug administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CellCept | Myfenax
Number analyzed (Participants) | 41 | 41
hours | 1.119 (0.7462) | 1.344 (1.1439)

8. Secondary Outcome: Summary of Participants With Adverse Events
Description: Summary of adverse events across three study time periods. The on-treatment time frame spanned the time during which study drug was administered. Relation to study drug was assessed by the investigator.
  The Adverse Event count includes serious and non-serious AEs. A serious AE (SAE) was any event that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity or congenital anomaly/birth defect or was an important medical event could have jeopardized the patient's safety or required medical or surgical intervention to prevent one of the outcomes listed above.
  Severity was measured on a three-point scale: mild, moderate, severe.
Time Frame: Day 1 up to Day 112
Population: Safety population. One participant discontinued the study prior to Period II so the Myfenax # participants analyzed is one less than the CellCept arm.
Measure: Number; unit: participants
Groups:
- CellCept: Participants experience while on CellCept during any of the three study periods. Doses of mycophenolate mofetil were at least 500 mg twice daily, morning and evening.
- Myfenax: Participants experience while on Myfenax during any of the three study periods. Doses of mycophenolate mofetil were at least 500 mg twice daily, morning and evening.
- Overall: Participant experience overall, i.e. all treatment experiences while on study are included
Arm/Group | CellCept | Myfenax | Overall
Number analyzed (Participants) | 43 | 42 | 43
participants
  Adverse Events | 15 | 17 | 26
  Related adverse events | 3 | 7 | 9
  Severe adverse events | 0 | 0 | 0
  Adverse events leading to discontinuation | 2 | 1 | 3
  Serious adverse events | 1 | 1 | 1
  Adverse events leading to death | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 112
Arm/Group | CellCept | Myfenax | Overall
Serious Adverse Events (participants affected / at risk) | 1/43 | 1/42 | 1/43
Other Adverse Events (participants affected / at risk) | 15/43 | 16/42 | 26/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CellCept (N=43) | Myfenax (N=42) | Overall (N=43)
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CellCept (N=43) | Myfenax (N=42) | Overall (N=43)
Diarrhoea (Gastrointestinal disorders) | 2 | 5 | 6
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 3
Nausea (Gastrointestinal disorders) | 0 | 2 | 2
Oedema peripheral (General disorders) | 2 | 0 | 2
Herpes simplex (Infections and infestations) | 2 | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 2
Blood pressure increased (Investigations) | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Headache (Nervous system disorders) | 1 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1
Periodontitis (Gastrointestinal disorders) | 1 | 0 | 1
Rectal discharge (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Application site erythema (General disorders) | 1 | 0 | 1
Chills (General disorders) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Blood triglycerides increased (Investigations) | 1 | 0 | 1
Cardiac murmur (Investigations) | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Bowenoid papulosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 1
Depression (Psychiatric disorders) | 1 | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
The study was designed to have a power of at least 80 % to show bioequivalence with 80 subjects. Only 43 subjects were included.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.